CLINICAL TRIAL: NCT06276686
Title: A Single Arm Feasibility Study of Exercise for Improving Long-course Chemoradiotherapy Efficacy in People With Locally Advanced Rectal Cancer
Brief Title: Exercise for Improving Long-course Chemoradiotherapy Efficacy in People With Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RS211 - 332296
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Rectal Carcinoma
Keywords: Exercise; chemoradiotherapy; Treatment efficacy; Locally advanced rectal cancer; Vigorous intensity aerobic interval exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm feasibility (Experimental): This study involves a single arm only. Therefore all consenting participants will receive the exercise intervention detailed in the protocol.
  The exercise interventions include an 11-week aerobic and resistance training delivered 2-weeks before chemoradiotherapy commences , in the 5-weeks of chemoradiotherapy and 4 weeks following chemoradiotherapy.
  2-days Aerobic exercise will be delivered on vigorous intensity on a cycle ergometer. This will be under the supervision of a trained physiotherapist. 2-days Resistance training will be home based with guidance of an exercise sheet.
  Interventions: Other: Supervised Vigorous intensity aerobic interval exercise

INTERVENTIONS:
Other: Supervised Vigorous intensity aerobic interval exercise — 11-weeks course of aerobic and resistance exercise, delivered 2 weeks before long course NACRT, 5-weeks during NACRT and 4 weeks post NACRT. Alongside twice weekly unsupervised resistance exercise training.
  Other Names: Unsupervised resistance exercise

SUMMARY:
This is a single arm feasibility study of exercise for improving long- course neoadjuvant chemoradiotherapy (NACRT) efficacy in people diagnosed with locally advanced rectal cancer. The study aims to recruit up to 30 patients from the Queen's Centre for Oncology and Haematology of Castle Hill Hospital, Cottingham, diagnosed with locally advanced rectal cancer. Consenting patients will be provided with an 11-week course of structured aerobic exercises and resistance training in the periods before, during and after their chemoradiotherapy treatment. The patients will be followed up for 6 months post long course neoadjuvant chemoradiotherapy (NACRT), with a total of 3 assessment periods.

DETAILED DESCRIPTION:
This study will take place at Castle Hill Hospital, where the participants' usual care will be given. The study will also recruit at this site. Patients, who have been diagnosed with locally advanced rectal cancer (LARC) long-course chemoradiotherapy (NACRT) will be pre-screened for any obvious exclusions with those that are potentially eligible approached by their clinical oncologist to discuss participation in these studies. If the patient is agreeable, further contact will be made by a member of the research team for further discussion. The aim is to include about 30 participants in this study. The participant information sheet will be provided and any uncertainties about the study raised by the potential participant will be addressed. The potential participant will be given sufficient time, up to a week, to consider their participation in the study, as typically, there is on average a 31-day period between decision to treat and start of neoadjuvant oncological treatment. After all questions are answered and provided the participant is willing to take part in the study, they will be asked to sign the consent form to confirm participation.

Once a participant agrees to taking part, their medical history, and investigations (performed as part of routine clinical care) will be reviewed. Each participant's data from investigational phase for rectal cancer up to long-course NACRT completion and re-assessment will be collected. Data on age, gender, stage of rectal cancer, and any comorbidities will be collected from medical notes. Participants will then be invited for a baseline assessment at Castle Hill Hospital in a designated risk assessed rehabilitation gym.

In this baseline assessment, further personal details will be taken from the patient, including height and weight measurements to calculate Body Mass Index (BMI), other descriptive information such as ethnicity will also be taken. The Patient Reported Outcome Measures (PROMs) will be completed either independently by participant or with the help of a member of the research team if required by participant. Some of the questionnaires, such as the EORTC-QLQ-CR29 and FACT-C, contained in this study contain some questions that may be perceived to be intrusive. They however are validated questionnaires that have previously been used in numerous rectal cancer research studies. To mitigate embarrassment, participants will be forewarned about the contents of these questionnaires and potential to cause embarrassment. Participants will be reminded that their response will be anonymised. Questions relating to stoma and sex life are presented much later in the questionnaires where rapport may have already been established. Participants will be encouraged to consult with their oncologist if the questionnaires prompt any treatment related problems they may be experiencing.

Participants will also on this day, be provided an accelerometer to wear on 7 randomly selected days at different timeframes of the study. Finally on this day an average of three resting heart rates will be taken. The value of the average of the resting hear rates will be used in calculating a heart rate reserve (HRR) of 60%, 70% and 80%. Using the formula (HRmax-RHR) × exercise intensity (60-80%) + RHR, where HRmax is 220-Age as found to be more effective in recent research. This will form one of the main bases for exercise intensity, to ensure individualisation of the supervised vigorous intensity interval training sessions.

The supervised hospital-based exercise will be delivered over an 11-week period. This is because long-course neoadjuvant chemoradiotherapy lasts 5-weeks. This design allows for a 2-week pre-neoadjuvant oncological and a 4-week post-neoadjuvant oncological treatment. Exercise will involve an hour long, twice weekly vigorous intensity aerobic interval exercise and twice weekly supported at-home resistance training for all 11-weeks of the study. Vigorous intensity aerobic interval exercise will be performed at 70-80% of heart rate reserve (HRR).

The first supervised vigorous intensity interval training class will feature an induction and orientation into the gym, facilities nearby, like a toilet and safety checks during exercise classes. Participants will be encouraged to be proactive in expressive their bodies response to the exercises and to seek help promptly if required. Participants will also on this day, be provided an accelerometer to wear on the days for unsupervised resistance training.

These supervised vigorous intensity interval training sessions will be delivered on an individual basis, lasting up to 60-minutes, performed on a cycle ergometer, and supervised by at least one trained exercise practitioner or a physiotherapist. The sessions will include a 5-minute warm up and 5-minute cool down. The interval phase will include up to 6 bouts of vigorous intensity interval training alternating between 5minutes of pedalling at up to 70-80% HRR and 2.5 minutes active rest, pedalling with no resistance at less than 60% HRR.

At the end of the exercise phase of the studies their will be a post-exercise assessment on the next working day of exercise completion, where all the information taken in the baseline assessment will be collected for comparison. Participants will not be seen again until their post-surgery phase, which will be 6 months from the start of NACRT. At this stage, information about Pathological complete response(PCR) or Radiological complete response (RCR) and tumour regression (TR) will be collected.

There will also be a semi-structured interview to explore participant satisfaction of the trial and acceptability of the exercises. Notes will be taken during the interview. The interview data will be coded and analysed via reflexive thematic analysis using the NVivo qualitative analysis software. People approached about the study in clinic who choose not to participant will be encouraged to discuss why they chose not to participate in a short survey with questions adapted from the study by Dwyer and colleagues in 2023. Information from this survey may be instrumental in adapting the study design appropriately to better serve this patient group.

There may be one additional research visit if sufficient data cannot be obtained from the medical notes. This will be face to face or via telephone, depending on participant preference and every attempt will be made to coordinate this with participants oncological appointment.

The total period of participation in the study for each patient will be at most 7 months, this is with a gap between completion of exercise and 6-month review from start of neoadjuvant oncological treatment. All research activities is planned to be completed within 18 months of receiving approval from the Research Ethics Committee(REC).

This study design will allow us to determine the proportion of people in our region with LARC who are willing to engage in structured outpatient exercise before, during and after long-course NACRT. There are not sufficient safety data in United Kingdom (UK) based subjects at present to justify incorporating exercise in all stages of the rectal cancer care pathway according to the current guidelines. Additionally, this study will also provide safety data by determining the proportion of LARC patients who are able to complete supervised vigorous Intensity Interval training and unsupervised training at home. The exploratory goals of these studies may provide indicative data on the impact of vigorous intensity training on quality of life and long-course NACRT efficacy.

Data generated from the study will be aggregated, anonymised, and used for publication in scientific journals and presented in abstract form at scientific meetings. All patient identifiable information will be always kept confidential. Anonymised data may be available to the scientific community following the end of the study. Data will be stored confidentially at the university of Hull for a maximum of 5 years for future research use if needed before it is fully destroyed. The management of the study will be overseen by the chief investigator. Regular meetings will be held by the chief investigator and members of the research team involved in the study to ensure all the correct steps are being taken and to address any issues that could exist.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have been diagnosed with locally advanced rectal cancer using MRI (Magnetic Resonance Imaging) and histological finding
* Have been offered long-course neoadjuvant chemoradiotherapy in the Queens Centre, Castle Hill Hospital
* Willing and able to comply with all study requirements
* Able and willing to voluntarily give informed consent to take part.

Exclusion Criteria:

* Inability to understand basic written and spoken English, as research materials will all be written in English.
* Any movement deficiencies limiting ability to engage in exercise.
* Impaired cognition and/or capacity limiting ability to provide informed consent.
* Cardiovascular and/or cardiopulmonary conditions that will impede ability to safely perform exercise.
* Severe psychiatric disorders.
* With any other health condition which oncologists and research team agrees will impede ability to safely perform exercises.
* Presence of metastatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | This will be monitored in the total 6months of participants engagement if the study
  The number of recruited participants/ total number of patients approached in percentage.
Attendance rate | This will be monitored in the total 6months of participants engagement if the study
  The number of supervised exercise sessions attended/ total number of available supervised exercise sessions in percentage.
withdrawal rate | This will be monitored in the total 6months of participants engagement if the study
  The number of participants who drop out of study/ total number of recruited participants in percentage.

SECONDARY OUTCOMES:
Serum Carcinoembryonic antigen levels | up to 4 weeks before neoadjuvant chemoradiotherapy (NACRT), immediately following chemoradiotherapy and 6-months following NACRT
  measuring Serum Carcinoembryonic antigen levels
FACT-C version 4 questionnaire for Quality of life | up to 4 weeks before NACRT, up to 1 week post NACRT and 6-months following NACRT
  measured using the FACT-C version 4 questionnaire
EORTC-QLQ-CR29 questionnaire for Quality of life | up to 4 weeks before NACRT, up to 1 week post NACRT and 6-months following NACRT
  measured using the EORTC-QLQ-CR29 questionnaire
Physical activity levels | up to 4 weeks before NACRT, up to 1 week post NACRT and 6-months following NACRT
  Using the 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: John Saxton, PhD, Study Chair — University of Hull
Locations (1):
- Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This falls outside the ethics approval obtained to conduct this study

REFERENCES:
- [Background] Chen T, Zhu H, Su Q. Effectiveness and Safety of Four Aerobic Exercise Intensity Prescription Techniques in Rehabilitation Training for Patients with Coronary Heart Disease. Cardiol Res Pract. 2022 Jul 15;2022:1647809. doi: 10.1155/2022/1647809. eCollection 2022. PMID 35874554
- [Background] Dwyer CP, Moses A, Rogers FM, Casey D, Joyce R, Hynes SM. A qualitative investigation of reasoning behind decisions to decline participation in a research intervention: A study-within-a-trial. J Health Psychol. 2023 Mar;28(4):374-387. doi: 10.1177/13591053211037736. Epub 2021 Aug 6. PMID 34355599
- [Background] Alejo LB, Pagola-Aldazabal I, Fiuza-Luces C, Huerga D, de Torres MV, Verdugo AS, Ortega Solano MJ, Felipe JL, Lucia A, Ruiz-Casado A. Exercise prehabilitation program for patients under neoadjuvant treatment for rectal cancer: A pilot study. J Cancer Res Ther. 2019 Jan-Mar;15(1):20-25. doi: 10.4103/jcrt.JCRT_30_17. PMID 30880749
- [Background] Loughney L, West MA, Moyses H, Bates A, Kemp GJ, Hawkins L, Varkonyi-Sepp J, Burke S, Barben CP, Calverley PM, Cox T, Palmer DH, Mythen MG, Grocott MPW, Jack S; Fit4Surgery group. The effects of neoadjuvant chemoradiotherapy and an in-hospital exercise training programme on physical fitness and quality of life in locally advanced rectal cancer patients: a randomised controlled trial (The EMPOWER Trial). Perioper Med (Lond). 2021 Jun 22;10(1):23. doi: 10.1186/s13741-021-00190-8. PMID 34154675
- [Background] Moug SJ, Mutrie N, Barry SJE, Mackay G, Steele RJC, Boachie C, Buchan C, Anderson AS. Prehabilitation is feasible in patients with rectal cancer undergoing neoadjuvant chemoradiotherapy and may minimize physical deterioration: results from the REx trial. Colorectal Dis. 2019 May;21(5):548-562. doi: 10.1111/codi.14560. Epub 2019 Feb 16. PMID 30657249